CLINICAL TRIAL: NCT00389974
Title: A Phase II Study of Sunitinib (SU11248; NSC 736511) an Oral Multi-Targeted Tyrosine Kinase Inhibitor, in Patients With Unresectable, Locally Advanced or Metastatic Cervical Carcinoma
Brief Title: Sunitinib Malate in Treating Patients With Uterine Cervical Cancer That is Stage IVB, Recurrent, or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00648; NCI-2014-00648 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCIC CTG IND.184; IND.184; NCIC-184 (Other: National Cancer Institute of Canada Clinical Trials Group); NCIC-184 (Other: CTEP)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2014-03

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Cell Carcinoma; Cervical Squamous Cell Carcinoma; Recurrent Cervical Cancer; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Sunitinib

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive sunitinib malate PO daily for 4 weeks. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or PR may receive 2 courses after CR or PR is reached.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial studies the side effects and how well sunitinib malate works in treating patients with cervical cancer which cannot be cured by standard therapy. Sunitinib malate may stop the growth of cervical cancer by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy (objective response rate) of sunitinib (sunitinib malate) given orally daily for 4 out of every 6 weeks in patients with unresectable, locally advanced or metastatic carcinoma of the cervix.

II. To assess the toxicity of sunitinib in patients with unresectable, locally advanced or metastatic carcinoma of the cervix.

III. To document time to progression, early objective progression rate, and, if objective responses are observed, response duration.

OUTLINE:

Patients receive sunitinib malate orally (PO) daily for 4 weeks. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) or partial response (PR) may receive 2 courses after CR or PR is reached.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell carcinoma or adenosquamous carcinoma of the cervix; patients with adenocarcinoma of the cervix will also be included since, although infrequent, their management in general is similar to those with squamous tumors
* Patients must have advanced (stage IVB) recurrent or persistent disease unsuitable for curative treatment by surgery and/or radiation therapy
* Presence of clinically and/or radiologically documented disease; at least one site of disease must be unidimensionally measurable as follows:

  * X-ray, physical exam >= 20 mm
  * Spiral computed tomography (CT) scan >= 10 mm
  * Non-spiral CT scan >= 20 mm
  * All radiology studies must be performed within 21 days prior to registration (within 28 days if negative)
* Patients must have a life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1; performance status (PS) 2 patients are eligible if, in the opinion of the investigator, they are suitable for inclusion in the study and are likely to be compliant with the study procedures (in particular the recommendations for supportive care and dose modifications)
* Patients may have had neoadjuvant or adjuvant chemotherapy
* Patients may have had concurrent chemoradiation; this is not considered neoadjuvant or adjuvant treatment
* Patients may have had no more than one prior chemotherapy regimen for recurrent metastatic disease; patients must be at least 28 days since last chemotherapy treatment and must have recovered from toxic effects
* Patients may have had prior radiation therapy, including external beam and/or intracavity radiation; a minimum of 28 days must have elapsed between the end of radiotherapy and registration onto the study; patients must have recovered from any acute toxic effects from radiation prior to registration; radiation must have involved < 30% of functioning bone marrow and there must be measurable disease outside the previously irradiated area (patients whose sole site of disease is in a previously irradiated area are ineligible UNLESS there is evidence of progression, or new lesions have been documented, in the irradiated field)
* Previous major surgery is permitted provided that it has been at least 28 days prior to patient registration and that wound healing has occurred
* Granulocytes (AGC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Bilirubin =< upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Calcium =< 3 mmol/L
* Serum creatinine =< ULN or creatinine clearance >= 60ml/min if creatinine is > ULN; creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by Cockcroft Formula
* Patient consent must be obtained according to local institutional and/or University Human Experimentation Committee requirements; it will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the National Cancer Institute of Canada (NCIC) Clinical Trials Group (CTG) study coordinator that such clearance has been obtained, before the trial can commence in that center; because of differing requirements, a standard consent form for the trial will not be provided; a copy of the initial full board Research Ethics Board (REB) approval and approved consent form must be sent to the central office; the patient must sign the consent form prior to randomization or registration; please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records
* Patients must be accessible for treatment, response assessment and follow-up; patients registered on this trial must be treated and followed at the participating center; this implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial; investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up
* In accordance with NCIC CTG policy, protocol treatment is to begin within 2 working days of patient registration; exceptions may be made however, regarding the washout period timing for prohibited medications

Exclusion Criteria:

* History of other malignancies, except: adequately treated non-melanoma skin cancer or other solid tumors curatively treated with no evidence of disease for >= 5 years
* Patients with known brain metastases; (a head CT is not necessary to rule out brain metastases, unless there is clinical suspicion of central nervous system [CNS] involvement); patients with known brain metastases will be excluded from this trial due to their poor prognosis and their likelihood of developing progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib
* Patients receiving concurrent treatment with other anti-cancer therapy or other investigational anticancer agents
* Patients who have received prior treatment with any other antiangiogenic agent or multi-targeted tyrosine kinase inhibitors (e.g., bevacizumab, sorafenib, pazopanib, thalidomide, AZD2171, AZD6474, AMG-706, PTK787, vascular endothelial growth factor [VEGF] Trap, etc.) are ineligible
* Corrected QT (QTc) prolongation (defined as a QTc interval equal to or greater than 500 msec) or other significant electrocardiogram (ECG) abnormalities; an ECG must be done within 14 days prior to registration
* Current or history of class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* Patients with prior anthracycline exposure, previous central thoracic radiation that included heart in radiation port, or a history of NYHA Class II cardiac function UNLESS

  * They are currently asymptomatic with respect to cardiac function AND
  * Left ventricular ejection fraction (LVEF) as assessed by multi gated acquisition (MUGA) at baseline is > lower limit of normal (LLN) of institution; the MUGA must be done within 14 days prior to registration
* Poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher)
* Myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
* History of pulmonary embolism within the past 12 months
* History of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
* Patients who require use of therapeutic doses of Coumadin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis; Note: low molecular weight heparin is permitted provided the patient's international normalized ratio (INR) is =< 1.5; INR must be done within 7 days prior to registration
* Patients with bowel obstruction or any condition (e.g. gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets
* Patients with serious illness or medical condition which would not permit the patient to be managed according to the protocol including, but not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements
  * Active uncontrolled infection
  * Any other medical conditions that might be aggravated by treatment
  * Serious or non-healing wound, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
* Use of agents with proarrhythmic potential (terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, and flecainide) is not permitted during the study
* Patients receiving azole antifungals (ketoconazole, itraconazole), clarithromycin, erythromycin, diltiazem, verapamil, human immunodeficiency virus (HIV) protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir) and delavirdine are not eligible unless >= 7 days since last dose before starting sunitinib and no dosing during the trial; patients receiving rifampin, rifabutin, carbamazepine, phenobarbital, phenytoin, St. John's wort, efavirenz and tipranavir are not eligible unless >= 12 days since last dose before starting sunitinib and no dosing during the trial
* Patients with pre-existing hypothyroidism prior to enrollment are ineligible unless they are euthyroid on medication
* Some women enrolled on this study will have had a prior hysterectomy for cervical cancer

  * Pregnant or lactating women; (N.B.: All women of childbearing potential must have a negative urine beta- human chorionic gonadotropin (beta-HCG) pregnancy test within 7 days prior to registration)
  * Women of childbearing potential who do not agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; (should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately)
* Known HIV-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Mackay, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sunitinib Malate)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated patients
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 44 [28 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (PR or CR)
Description: It is defined as per the Response Evaluation Criteria In Solid Tumors criteria for at least 4 weeks. The 95% confidence interval for response rate will be calculated.
Time Frame: Up to 2 years
Population: All patients evaluable for response
Measure: Number (95% Confidence Interval); unit: percentage of evalubale patients
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 19
percentage of evalubale patients | 0 [0 to 17.6]

ADVERSE EVENTS:
Arm/Group | Treatment (Sunitinib Malate)
Serious Adverse Events (participants affected / at risk) | 14/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sunitinib Malate) (N=19)
Hospitalization for Pain-Pelvis (General disorders) | 1
Fistula (Gastrointestinal disorders) | 1
Urinary obstruction (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal Obstruction (Renal and urinary disorders) | 1
Hospitalization for Bowel Obstruction (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Function Liver Tests (Investigations) | 1
Hospitalization for Rectovaginal Fistula (Renal and urinary disorders) | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Hemorrhage: vagina (Blood and lymphatic system disorders) | 1
Chest Pain (General disorders) | 1
Pelvic Pain (General disorders) | 1
Periorbital Edema (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sunitinib Malate) (N=19)
Auditory/Ear - Other (Ear and labyrinth disorders) | 2
Supraventricular arrhythmia Sinus tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 10
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Fatigue (General disorders) | 17
Insomnia (General disorders) | 8
Patient odor (General disorders) | 1
Rigors/chills (General disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Bruising (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hand-foot (Skin and subcutaneous tissue disorders) | 5
Hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Induration (Skin and subcutaneous tissue disorders) | 2
Nail changes (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 8
Urticaria (Skin and subcutaneous tissue disorders) | 1
Dermatology - Other (yellowing of the skin) (Skin and subcutaneous tissue disorders) | 10
Hot flashes (Endocrine disorders) | 4
Anorexia (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 15
Distension (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 4
Enteritis (Gastrointestinal disorders) | 1
Fistula, GI Rectum (Gastrointestinal disorders) | 1
Fistula, GI Small bowel NOS (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 12
Hemorrhoids (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Mucositis (clinical exam) Oral cavity (Gastrointestinal disorders) | 10
Mucositis (functional/symptomatic) Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Taste alteration (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 10
GI - Other (Gastrointestinal disorders) | 6
Hemorrhage pulmonary Nose (Blood and lymphatic system disorders) | 4
Hemorrhage, GI Anus (Blood and lymphatic system disorders) | 1
Hemorrhage, GI Lower GI NOS (Blood and lymphatic system disorders) | 1
Hemorrhage, GI Oral cavity (Blood and lymphatic system disorders) | 1
Hemorrhage, GI Rectum (Blood and lymphatic system disorders) | 3
Hemorrhage, GU Bladder (Blood and lymphatic system disorders) | 2
Hemorrhage, GU Urinary NOS (Blood and lymphatic system disorders) | 2
Hemorrhage, GU Vagina (Blood and lymphatic system disorders) | 7
Infection with normal ANC Abdomen NOS (Infections and infestations) | 1
Infection with normal ANC Bladder (Infections and infestations) | 1
Infection with normal ANC Dental-tooth (Infections and infestations) | 1
Infection with normal ANC Skin (Infections and infestations) | 1
Iinfection with normal ANC Urinary tract NOS (Infections and infestations) | 1
Infection with unknown ANC Bladder (Infections and infestations) | 1
Infection with unknown ANC Vagina (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 1
Edema: head and neck (Blood and lymphatic system disorders) | 4
Edema: limb (Blood and lymphatic system disorders) | 7
Edema: trunk/genital (Blood and lymphatic system disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Mood alteration Agitation (Nervous system disorders) | 1
Mood alteration Anxiety (Nervous system disorders) | 3
Mood alteration Depression (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 3
Watery eye (Eye disorders) | 1
Ocular - Other (Eye disorders) | 1
Pain Abdomen NOS (General disorders) | 10
Pain Back (General disorders) | 10
Pain Bladder (General disorders) | 1
Pain Bone (General disorders) | 2
Pain Chest/thorax NOS (General disorders) | 4
Pain Extremity-limb (General disorders) | 5
Pain Head/headache (General disorders) | 8
Pain Joint (General disorders) | 2
Pain Lip (General disorders) | 1
Pain Muscle (General disorders) | 2
Pain Neck (General disorders) | 1
Pain Oral cavity (General disorders) | 2
Pain Pelvis (General disorders) | 7
Pain Rectum (General disorders) | 1
Pain Throat/pharynx/larynx (General disorders) | 3
Pain Tumour pain (General disorders) | 1
Pain Urethra (General disorders) | 2
Pain Vagina (General disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Voice changes (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 2
Bladder spasms (Renal and urinary disorders) | 1
Fistula, GU Bladder (Renal and urinary disorders) | 1
Fistula, GU Vagina (Renal and urinary disorders) | 1
Leak, GU Urethra (Renal and urinary disorders) | 1
Obstruction, GU Urethra (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less